CLINICAL TRIAL: NCT04262193
Title: Dual-Orexin Antagonism As a Mechanism for Improving Sleep and Drug Abstinence in Opioid Use Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not meet enrollment goals.
Sponsor: Wayne State University (Other)
Collaborators: Henry Ford Health System (Other); Ascension Brighton Center for Recovery (Unknown)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor of Psychiatry and Behavioral Neurosciences; and Director, Substance Abuse Research Division, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DORA, Sleep and Opioid Use
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Opioid-use Disorder; Sleep
MeSH Terms: conditions — Opioid-Related Disorders | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the 2 parallel groups for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Suvorexant (20mg) and placebo research tablets will appear identical.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Suvorexant placebo (Placebo Comparator): Placebo (inert) tablet
  Interventions: Drug: Suvorexant Placebo
- Suvorexant 20mg (Experimental): Suvorexant 20mg tablet
  Interventions: Drug: Suvorexant

INTERVENTIONS:
Drug: Suvorexant — In each group, the participant will take 1 tablet (placebo or 20mg) 30 minutes before bedtime.
  Other Names: Belsomra
  Arms: Suvorexant 20mg
Drug: Suvorexant Placebo — Suvorexant Placebo
  Arms: Suvorexant placebo

SUMMARY:
Summary of Study Protocol. This project is designed to test neurobehavioral mechanisms underlying effects of the dual orexin-1/2 receptor antagonist suvorexant on sleep efficiency and opioid abstinence, and whether these outcomes are independent of one another. This will be the first study to investigate whether suvorexant improves outpatient opioid abstinence and sleep efficiency; and whether improving sleep mediates the improved opioid abstinence outcome. 120 participants with opioid use disorder (OUD) will complete this intent-to-treat study.

DETAILED DESCRIPTION:
Study Design. Using a placebo-controlled, parallel-group, randomized clinical trial design, we will prospectively evaluate whether nightly treatment with the orexin-1/2 receptor antagonist suvorexant (20 mg/day PO), relative to placebo, can increase outpatient opioid abstinence and improve sleep efficiency (sleep time per time-in-bed) as a mediator/moderator among patients with OUD. We include current medication for treating OUD, as well as treatment site, as stratification factors in the group allocation. Using power and sample size calculations, we estimate that 120 participants will suffice to test our hypotheses.

The study aims to test three co-primary hypotheses:

Hypothesis 1: Relative to placebo, suvorexant (20 mg/day) will significantly increase percentage opioid abstinence during outpatient weeks 1-13.

Hypothesis 2: Relative to placebo, suvorexant will improve sleep efficiency.

Hypothesis 3: Higher inpatient sleep efficiency will be associated with increased outpatient opioid abstinence (independent of experimental group assignment).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* Males and non-pregnant females who agree to medically accepted birth control for the duration of the study
* Meet DSM-5 criteria for opioid use disorder (any severity level) alone or comorbid with stable medical diseases (except for certain medications [see below])

Exclusion Criteria:

* Body mass index >38
* Acute/unstable illness: conditions making it unsafe for participation, conditions with potential to disturb sleep (i.e. acute pain, respiratory infection)
* Chronic illnesses; renal failure, liver disease, seizures, and dementing illnesses
* Current psychiatric disease: psychosis, bipolar disorder, PTSD
* Smoking during the night (11pm-7am). Nicotine replacement therapy is allowed
* Medications including anxiolytics, hypnotics (both prescription and OTC), sedating antidepressants, anticonvulsants, sedating H1 antihistamines (non-sedating second generation H4 antihistamines are allowed), systemic steroids, respiratory stimulants and decongestants, prescription and OTC stimulants, prescription and OTC diet aids, herbal preparations, and narcotic analgesics. All medications and doses will be documented
* Sleep-disordered breathing and periodic leg movements (PLMs) defined as ≥ 10 apnea-hypopneas or PLM events related to EEG arousal per hour of sleep time, or any other primary sleep (e.g. narcolepsy, restless legs syndrome) or circadian disorder
* Night-shift work, which would alter circadian rhythm and be a confound in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Opioid abstinence | up to 13 weeks
  Percentage of opioid-free urine drug screens (UDS)
Sleep efficiency | Sleep efficiency is measured on the evening of the first medication dose
  Sleep efficiency equals sleep time (determined by standardized scoring of electroencephalogram recordings) divided by time in bed

SECONDARY OUTCOMES:
Daily sleep questionnaire | Change in sleep quality scores from inpatient stay to outpatient weeks 2, 6 and 10
  Morning (post-awakening) assessment of sleep quality
Actigraphic assessment of sleep | Change in total activity counts across outpatient weeks 2, 6 and 10
  Actigraphic assessment of motion (activity counts), measured with Actiwatch and scoring software; motion is absent during sleep.
Weekly sleep questionnaire | Change in sleep quality scores across outpatient weeks 1, 4, 8 and 12
  Retrospective (past-week) self-report of sleep quality on each of 4 outpatient weeks
Timeline followback interview assessment of substance use | Once weekly (in conjunction with urine drug screen) on outpatient weeks 1 through 13
  Percentage of outpatient weeks with substance use (opioids, methadone, buprenorphine, cocaine metabolites, benzodiazepines, barbiturates, cannabinoids, amphetamines)
Urinary cortisol | Measured at 11pm on nights 4, 6, 8 (coordinated with sleep efficiency and melatonin assessments) and the following day (7am and 3pm on days 5, 7, 9) on the inpatient unit
  Change in cortisol levels in picogram per milliliter (pg/ml) across 24 hour interval used to measure circadian rhythm
Urinary melatonin | Measured at 11pm on nights 4, 6, 8 (coordinated with sleep efficiency and cortisol assessments) and the following day (7am and 3pm on days 5, 7, 9) on the inpatient unit
  Change in melatonin levels in picograms per milliliter (pg/ml) across 24 hour interval used to measure circadian rhythm
Clinical Global Impression (CGI) | Change in CGI subscale scores across outpatient weeks 4, 8, and 12
  CGI subscale scores for improvement and severity. Each subscale is scored on a 1-7 scale. Higher scores indicate worse (more severe) outcomes.
Short Form-36 v2 Health Survey | Change in overall health total score across outpatient weeks 4, 8, and 12
  Overall health assessment. The 36 items are grouped into 8 dimensions: physical functioning, physical and emotional limitations, social functioning, bodily pain, general and mental health. Each scale is directly transformed into a 0-100 scale. Lower scores on each scale indicate greater disability.
Medication satisfaction | Change in medication satisfaction score across outpatient weeks 4, 8, and 12
  Assessment of satisfaction with assigned medication condition, on 1-7 Likert scale. Higher scores indicate greater medication satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
This plan is under development. This project was funded under the NIH HEAL Initiative, which requires data sharing through a repository; IPD details are being determined.
Supporting Information: Study Protocol
Time Frame: Electronic copies of publications will be deposited within 4 weeks of acceptance. Underlying primary data will be made publicly available as soon as possible (time frame to be determined).
Access Criteria: De-identified data (still being processed) will be placed in the NSRR (National Sleep Research Resource) repository.
URL: https://sleepdata.org/